CLINICAL TRIAL: NCT05596981
Title: The Gut Microbiome Changes in FMS-like Tyrosine Kinase 3 (FLT3)-ITD Positive Acute Myeloid Leukemia Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation With or Without Sorafenib Maintenance Post-transplantation
Brief Title: The Gut Microbiome in FLT3-ITD+ AML Undergoing Allo-HSCT With Or Without Sorafenib Maintenance After Allo-HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Xuanli, professor, Nanfang Hospital, Southern Medical University
Other Study IDs: Microbiota-Sora-FLT3+AML-2022
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation; Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Hematopoietic Stem Cell Transplantation; Gut Microbiome; Sorafenib; Acute Myeloid Leukemia; FLT3-ITD
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, bone marrow and/or peripheral blood samples will be collected on the first day of regimen therapy for allo-HSCT, then subsequently every 28 days until discharging from the hospital, whichever occurs sooner. After discharging from the hospital, specimens will continuously be collected on the day before sorafenib maintenance therapy, then subsequently every 28 days until 3 months after receiving sorafenib maintenance therapy. The samples were tagged and stored at -80°C until retrieval for DNA extraction and cytokine detection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sorafenib group: FLT3-ITD+ AML patients who receive sorafenib maintenance therapy after Allo-HSCT. Sorafenib will be used from day 30 to 180 post-transplantation. The initial dose of sorafenib is 400 mg orally twice daily and is adjusted in case of suspected toxicity or resistance (dose range, 200-800 mg daily).
  Interventions: Drug: Sorafenib
- non-sorafenib group: FLT3-ITD+ AML patients who do not receive sorafenib maintenance therapy after Allo-HSCT.

INTERVENTIONS:
Drug: Sorafenib — The initial dose of sorafenib is 400 mg orally twice daily and is adjusted in case of suspected toxicity or resistance (dose range, 200-800 mg daily).
  Other Names: Nexavar; BAY 43-9006; BAY-673472; BAY 545-9085
  Groups: sorafenib group

SUMMARY:
This prospective trial investigates the effect of sorafenib maintenance therapy in FLT3-ITD AML patients after allo-HSCT in terms of gut microbiome.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is used as a potentially curative therapy for patients with hematopoietic malignancies. Sorafenib, an inhibitor of multiple kinases including FLT3, has shown promising activity in FLT3-ITD-positive AML. Our previous studies demonstrated that sorafenib maintenance post-transplantation could improve the outcomes of FLT3-ITD-positive AML patients, which is associated with sorafenib enhancing the graft-versus-leukemia (GVL) effect. Recent studies show that gut microbiome is associated with graft-versus-host-disease (GVHD) and GVL. However, the exact mechanism of sorafenib enhancing the GVL effect and the influence of gut microbiome on sorafenib maintenance after allo-HSCT remain unknown.

ELIGIBILITY:
Inclusion Criteria:

* FLT3-ITD Positive AML
* Allo-HSCT Recipients

Exclusion Criteria:

* Intolerance to sorafenib pre-transplantation
* Cardiac dysfunction (particularly congestive heart failure)
* Hepatic abnormalities (bilirubin ≥ 3 mg/dL, aminotransferase> 2 times the upper limit of normal)
* Renal dysfunction (creatinine clearance rate < 30 mL/min)
* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (according to the investigators' decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FLT3-ITD Positive AML Undergoing Allo-HSCT
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Variation of Gut Microbiota Composition and Diversity | 3 months
  Variation of gut microbiota composition and diversity, as determined by 16s rRNA sequencing of serial stool samples, during Sorafenib Maintenance Therapy.

SECONDARY OUTCOMES:
Variation of gut barrier integrity | 3 months
  As determined by serum levels of zonulin, I-FABP, and citrulline or other potential candidates.
NRM | 1 year
  Non-relapse mortality (NRM)
Acute GVHD | 100 days
  Acute Graft-Versus-Host-Disease
Chronic GVHD | 1 year
  Chronic Graft-Versus-Host-Disease
AEs | 1 year
  Adverse Events
OS | 1 year
  Overall survival
LFS | 1 year
  Leukemia-free survival
Relapse | 1year
  Cumulative incidence of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Li Xuan, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sidaway P. Intestinal microbiota predict HSCT outcome. Nat Rev Clin Oncol. 2020 May;17(5):275. doi: 10.1038/s41571-020-0351-9. No abstract available. PMID 32203272
- [Background] Spencer CN, McQuade JL, Gopalakrishnan V, McCulloch JA, Vetizou M, Cogdill AP, Khan MAW, Zhang X, White MG, Peterson CB, Wong MC, Morad G, Rodgers T, Badger JH, Helmink BA, Andrews MC, Rodrigues RR, Morgun A, Kim YS, Roszik J, Hoffman KL, Zheng J, Zhou Y, Medik YB, Kahn LM, Johnson S, Hudgens CW, Wani K, Gaudreau PO, Harris AL, Jamal MA, Baruch EN, Perez-Guijarro E, Day CP, Merlino G, Pazdrak B, Lochmann BS, Szczepaniak-Sloane RA, Arora R, Anderson J, Zobniw CM, Posada E, Sirmans E, Simon J, Haydu LE, Burton EM, Wang L, Dang M, Clise-Dwyer K, Schneider S, Chapman T, Anang NAS, Duncan S, Toker J, Malke JC, Glitza IC, Amaria RN, Tawbi HA, Diab A, Wong MK, Patel SP, Woodman SE, Davies MA, Ross MI, Gershenwald JE, Lee JE, Hwu P, Jensen V, Samuels Y, Straussman R, Ajami NJ, Nelson KC, Nezi L, Petrosino JF, Futreal PA, Lazar AJ, Hu J, Jenq RR, Tetzlaff MT, Yan Y, Garrett WS, Huttenhower C, Sharma P, Watowich SS, Allison JP, Cohen L, Trinchieri G, Daniel CR, Wargo JA. Dietary fiber and probiotics influence the gut microbiome and melanoma immunotherapy response. Science. 2021 Dec 24;374(6575):1632-1640. doi: 10.1126/science.aaz7015. Epub 2021 Dec 23. PMID 34941392
- [Background] Peled JU, Gomes ALC, Devlin SM, Littmann ER, Taur Y, Sung AD, Weber D, Hashimoto D, Slingerland AE, Slingerland JB, Maloy M, Clurman AG, Stein-Thoeringer CK, Markey KA, Docampo MD, Burgos da Silva M, Khan N, Gessner A, Messina JA, Romero K, Lew MV, Bush A, Bohannon L, Brereton DG, Fontana E, Amoretti LA, Wright RJ, Armijo GK, Shono Y, Sanchez-Escamilla M, Castillo Flores N, Alarcon Tomas A, Lin RJ, Yanez San Segundo L, Shah GL, Cho C, Scordo M, Politikos I, Hayasaka K, Hasegawa Y, Gyurkocza B, Ponce DM, Barker JN, Perales MA, Giralt SA, Jenq RR, Teshima T, Chao NJ, Holler E, Xavier JB, Pamer EG, van den Brink MRM. Microbiota as Predictor of Mortality in Allogeneic Hematopoietic-Cell Transplantation. N Engl J Med. 2020 Feb 27;382(9):822-834. doi: 10.1056/NEJMoa1900623. PMID 32101664
- [Background] Han L, Zhao K, Li Y, Han H, Zhou L, Ma P, Fan Z, Sun H, Jin H, Jiang Z, Liu Q, Peng J. A gut microbiota score predicting acute graft-versus-host disease following myeloablative allogeneic hematopoietic stem cell transplantation. Am J Transplant. 2020 Apr;20(4):1014-1027. doi: 10.1111/ajt.15654. Epub 2019 Dec 12. PMID 31605563
- [Background] Andrews MC, Duong CPM, Gopalakrishnan V, Iebba V, Chen WS, Derosa L, Khan MAW, Cogdill AP, White MG, Wong MC, Ferrere G, Fluckiger A, Roberti MP, Opolon P, Alou MT, Yonekura S, Roh W, Spencer CN, Curbelo IF, Vence L, Reuben A, Johnson S, Arora R, Morad G, Lastrapes M, Baruch EN, Little L, Gumbs C, Cooper ZA, Prieto PA, Wani K, Lazar AJ, Tetzlaff MT, Hudgens CW, Callahan MK, Adamow M, Postow MA, Ariyan CE, Gaudreau PO, Nezi L, Raoult D, Mihalcioiu C, Elkrief A, Pezo RC, Haydu LE, Simon JM, Tawbi HA, McQuade J, Hwu P, Hwu WJ, Amaria RN, Burton EM, Woodman SE, Watowich S, Diab A, Patel SP, Glitza IC, Wong MK, Zhao L, Zhang J, Ajami NJ, Petrosino J, Jenq RR, Davies MA, Gershenwald JE, Futreal PA, Sharma P, Allison JP, Routy B, Zitvogel L, Wargo JA. Gut microbiota signatures are associated with toxicity to combined CTLA-4 and PD-1 blockade. Nat Med. 2021 Aug;27(8):1432-1441. doi: 10.1038/s41591-021-01406-6. Epub 2021 Jul 8. PMID 34239137
- [Background] Peled JU, Devlin SM, Staffas A, Lumish M, Khanin R, Littmann ER, Ling L, Kosuri S, Maloy M, Slingerland JB, Ahr KF, Porosnicu Rodriguez KA, Shono Y, Slingerland AE, Docampo MD, Sung AD, Weber D, Alousi AM, Gyurkocza B, Ponce DM, Barker JN, Perales MA, Giralt SA, Taur Y, Pamer EG, Jenq RR, van den Brink MRM. Intestinal Microbiota and Relapse After Hematopoietic-Cell Transplantation. J Clin Oncol. 2017 May 20;35(15):1650-1659. doi: 10.1200/JCO.2016.70.3348. Epub 2017 Mar 15. PMID 28296584